CLINICAL TRIAL: NCT06062641
Title: Selinexor Combined With R-GDP Regimen for TP53-altered Relapsed/Refractory Diffuse Large B-cell Lymphoma: a Single Arm, Single Center, Phase II Study
Brief Title: Selinexor Combined With R-GDP Regimen for TP53-altered R/R DLBCL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Vice president，Ruijin hospital, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-XLYM-002
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Relapsed or Refractory B-cell Lymphoma
Keywords: TP53-altered; Relapsed/Refractory; Diffuse Large B Cell Lymphoma; Selinexor
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SR-GDP (Experimental)
  Interventions: Drug: SR-GDP

INTERVENTIONS:
Drug: SR-GDP — Selinexor 40mg/d，po d1,8,15; rituximab 375mg/m2, iv d1; gemcitabine 1g/m2, iv d1,8; cisplatin 25mg/m2, iv d1-3; dexamethasone 40mg，po/iv d1-4 (If patient>70y, the dosage should be changed to 20mg). Each cycle lasts for 21 days, with a maximum of 6 cycles of combination therapy. For patients who achieved PR or better response at the end of combination therapy, they will start receiving single-agent selinexor 40mg treatment (qw) in cycles of 28 days until disease progression (PD) or unacceptable toxicity occurs.

SUMMARY:
To evaluate the efficacy and safety of selinexor combined with R-GDP regimen in the treatment of patients with TP53-altered relapsed or refractory B-cell lymphoma.

DETAILED DESCRIPTION:
This study is a single-arm, open-label exploratory clinical trial. To evaluate the efficacy and safety of selinexor combined with R-GDP regimen in the treatment of patients with TP53-altered relapsed or refractory B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18
2. Pathologically confirmed primary DLBCL or previously diagnosed indolent lymphoma (e.g., follicular lymphoma) transformation to DLBCL with TP53 deletion or mutation confirmed by FISH or next-generation sequencing.
3. Received at least 1 but no more than 3 previous lines of systemic therapy for DLBCL, and was relapsed or refractory to the last line of therapy Salvage chemoimmunotherapy and subsequent stem cell transplantation are considered the same first-line systemic therapy Maintenance therapy will not be counted separately as first-line systemic therapy Radiotherapy for curative treatment of localized DLBCL lesions does not count as first-line systemic therapy
4. Presence of measurable positron-emission tomography (PET) -positive lesions with at least one lymph node lesion long diameter (LDi) > 1.5 cm or an extra-nodal lesion LDi > 1 cm (according to the Lugano classification, 2014 version)
5. Bone marrow function was good at screening Absolute neutrophil count (ANC) ≥1×109/L Platelet count ≥50×109/L (no platelet transfusion < 14 days before cycle 1 day 1, C1D1) Hemoglobin ≥8.0 g/dL (no red blood cell transfusion < 14 days before C1D1)
6. Good liver and kidney function, namely:

   AST or ALT ≤2.5× upper normal value limit (ULN), or ≤5×ULN in the presence of known lymphoma involving the liver Serum total bilirubin ≤2×ULN, or when Gilbert's syndrome or known lymphoma involves the liver≤5×ULN CrCl≥30 mL/min according to the Cockcroft-Gault formula
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤2
8. Estimated life expectancy at screening was > 3 months
9. Agree to use a highly effective contraceptive during the study, which lasts for 12 months after the last dose of study treatment

Exclusion Criteria:

* Patients who met any of the following exclusion criteria were not eligible for the study:

  1. Prior treatment with selinexor or another XPO1 inhibitor
  2. There are contraindications to any drug in the combination therapy
  3. Receipt of any standard or investigational anti-DLBCL therapy <21 days before C1D1 (including non-palliative radiotherapy, chemotherapy, immunotherapy, radioimmunotherapy, or any other anticancer therapy) (Palliative radiotherapy for non-target lesions was allowed)
  4. Undergone major surgery <14 days before C1D1
  5. Hematopoietic stem cell transplantation /CAR-T therapy requirements are as follows:

     Autologous hematopoietic stem cell transplantation (HSCT) <100 days or allogeneic HSCT <180 days prior to C1D1 Active graft-versus-host disease (GVHD) after allogeneic HSCT (or inability to discontinue GVHD therapy or preventive therapy) CAR-T cell infusion <90 days before cycle 1
  6. Presence of grade ≥2 neuropathy (CTCAE, v.5.0)
  7. Presence of any life-threatening disease, medical condition, or organ system dysfunction that is considered by the investigator to be likely affecting patient safety or adherence to study procedures
  8. Uncontrolled (i.e., clinically unstable) infection within 7 days before the first dose of study treatment and required treatment with intravenous antibiotics, antiviral drugs or antifungal drugs; However, prophylactic use of these agents was allowed.
  9. Patients with active HBV, HCV, or HIV infection. Participants who were HBsAg positive and/or HBcAb positive but HBV-DNA negative, and/or HCV antibody positive but HCV-RNA negative were allowed to participate (the upper limit of normal values for HBV-DNA and HCV-RNA were based on the values available at each participating center).
  10. Inability to swallow tablets, presence of a malabsorption syndrome, or any other condition that may interfere with absorption of the study drug
  11. Lactating or pregnant women
  12. Unable or unwilling to sign the ICF
  13. Patients who were considered by the investigator to be significantly below tolerable weight
  14. Patients who received live attenuated vaccine within 28 days prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | At the end of Cycle 6 (each cycle is 21 days)
  Objective Response Rate (ORR) : The investigator-assessed best disease status of patients with TP53-altered R/R DLBCL was the rate of Complete Response (CR) or Partial Response (PR)

SECONDARY OUTCOMES:
progression free survival | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of diagnosis until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria,or death from any cause, whichever occurred first.
overall survival | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of diagnosis to the date of death from any cause. Reported is the percentage of participants with event. of disease progression or relapse, using 2014 Lugano criteria,or death from any cause, whichever occurred first.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Up to 30 days after completion of study treatment
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, PhD, MD, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanhai, China

IPD SHARING:
Plan to Share IPD: No